CLINICAL TRIAL: NCT00606541
Title: An Open Label, Double-blind Discontinuation Study of Quetiapine (Extended Release) XR in Social Anxiety Disorder
Brief Title: An Open Label, Double-blind Discontinuation Study of Quetiapine Extended Release(XR)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was terminated by the sponsor due to budgetary issues
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00002146; eIRB2146; IRUSQUET0452
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2012-12

CONDITIONS: Social Anxiety Disorder
Keywords: Social Anxiety Disorder; Quetiapine XR; Prevention; tolerability
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Quetiapine XR 50mg-400mg per day
  Interventions: Drug: Quetiapine XR
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine XR — This is an investigator-initiated, single site study, consisting of two phases: 1) 8-week, open label treatment with quetiapine XR (50-400 mg/day) in subjects (n=55 in order to randomize 20 into each of the quetiapine XR and PBO arms in the 2nd phase of the study) with SAD; and 2) in those who demonstrate at least minimal improvement (i.e. CGI≤3), 12-weeks randomized, double-blind treatment with either quetiapine XR or placebo (PBO).
  Other Names: Seroquel XR
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Purpose of Study: To examine 1) the short and long-term effectiveness and tolerability of quetiapine (extended release) XR for the treatment of social anxiety disorder (SAD); and 2) continuation effects of quetiapine XR in preventing SAD relapse.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* A primary diagnosis of SAD,using Diagnostic Standard Manual IV(DSM-IV) criteria
* Minimum CGI severity score of 4 and minimum Brief Social Phobia Scale (BSPS) score of 20 at baseline
* Written informed consent
* A negative serum pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, mental retardation or other pervasive developmental disorder, or cognitive disorder due to a general medical condition
* Any current primary anxiety disorder other than SAD or current primary depression
* History of substance abuse or dependence within the last 6 months
* Suicide risk or serious suicide attempt within the last year
* Clinically significant medical condition or laboratory abnormality
* Women of childbearing potential who are unwilling to practice an acceptable method of contraception
* Subjects needing concurrent use of psychotropic medications
* History of hypersensitivity to quetiapine
* History of cataracts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Kaplan Meier survival of Clinical Global Impression of Improvement (CGI-I) | 20 weeks

SECONDARY OUTCOMES:
Percentage of CGI-I, BSPS, SPIN | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States